CLINICAL TRIAL: NCT00500565
Title: Randomized, Double Blind, Controlled Trial of Two Methods of Postoperative Pain Management Following Free Transverse Rectus Abdominous Musculocutaneous (TRAM) Flap for Breast Reconstruction
Brief Title: Pain Management Following TRAM Flap for Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: I-Flow (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID03-0046
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; On-Q Pain Relief System; Transverse Rectus Abdominous Myocutaneous; Breast Reconstruction; TRAM flap; Bupivicaine; Pain Management
MeSH Terms: conditions — Breast Neoplasms; Agnosia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- On-Q pump with Saline (Experimental): On-Q Pump with Saline
  Interventions: Drug: Saline
- On-Q Pump with Bupivicaine (Experimental): On-Q Pump with bupivicaine
  Interventions: Drug: Bupivicaine

INTERVENTIONS:
Drug: Saline — On-Q Pain Pump filled with Saline. The On-Q pump will be connected to the catheter to deliver a constant flow of saline for up to 5 days.
  Arms: On-Q pump with Saline
Drug: Bupivicaine — On-Q Pain Pump filled with 0.375% Bupivicaine through two catheters at a total rate of 4 cc/hr over 111 hours. The On-Q pump will be connected to the catheter to deliver a constant flow of Bupivicaine for up to 5 days.
  Arms: On-Q Pump with Bupivicaine

SUMMARY:
The objective of this pilot study is to examine the efficacy of the ON~Q Pain Relief System plus Intravenous Patient Controlled Analgesia (IVPCA) with Morphine vs IV PCA alone in patients undergoing free transverse rectus abdominis musculocutaneous (TRAM) flap surgery. The primary outcome measure will be postoperative opioid analgesia requirements. Other outcomes will also be assessed, including pain scores, quality of recovery, and resource utilization.

DETAILED DESCRIPTION:
Inadequate control of surgical pain after free TRAM procedures may lead to complications and delay recovery time. This could lead to a longer stay in the hospital. The standard care for pain after a free TRAM procedure has been with drugs that are anesthetics. Unfortunately, these anesthetics are not long lasting and usually require the use of opioids (morphine or hydromorphone) to control "break-through" pain. A continuous delivery of local anesthetic to the wound site may provide better control of pain and decrease the need for the use of opioids. This may decrease the length of the hospital stay as well as other side effects associated with the treatment of pain.

Before the study, you will be asked questions about your health, your age, and about any allergies you may have. Women who are able to have children must have a negative blood pregnancy test. You will have already been scheduled to undergo a free TRAM flap procedure.

During free TRAM flap procedure, you will have two "soaker catheters" placed by the surgeon directly into the surgical site. The catheters are flexible tubes which will allow pain medicine (or saline) to be delivered directly to the donor wound site which is the abdominal site from where the tissue for breast reconstruction is taken. A small pump (On-Q pump) will be connected to the catheter to deliver a constant flow of pain medicine (or saline) for up to 5 days. The On-Q pump is completely portable and can be attached to your hospital gown to allow for movement.

You will be randomly assigned (as in the toss of a coin) to one of two groups. Participants in the first group will have the On-Q pump filled with saline. Participants in the other group will have the On-Q pump filled with bupivicaine.

Participants in both groups will receive IVPCA, which is the standard of care for pain relief. The IVPCA will be placed on PRN mode which means you will be able to press a button to deliver pain medication whenever you feel pain.

You will be asked questions about your pain and your recovery process every 6 hours while you are awake for up to 5 days. You will also be asked to fill out a questionnaire about pain once a day during treatment. It should take around 10 minutes to complete the questionnaire.

The catheters will be removed after 5 days of treatment (or your last day in the hospital, whichever is sooner) by one of the surgeons that participated in the surgery

During the study, if you experience any intolerable side effects or your doctor feels it is in your best interest to stop treatment, you will be taken off the study and other treatment options will be discussed with you.

This is an investigational study. The On-Q device, PCA, and bupivicaine are FDA approved and commercially available. Up to 60 participants will take part in this study (30 in each group). All will be enrolled at The University of Texas (UT) MD Anderson Cancer Center (MDACC).

This protocol is partially funded by a research grant from the I-Flow Corporation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with or undergoing unilateral elective free TRAM flap for breast reconstruction, immediate or delayed, with or without a surgical revision of the contralateral breast for asymmetry.
* American Society of Anesthesiology Physical Status I - III patients.
* Patients has given voluntary written informed consent before performance of any study-related procedure.

Exclusion Criteria:

* Patients undergoing bilateral TRAM flap reconstruction.
* Patients with a prior allergic reaction to Marcaine (bupivacaine) or other amide local anesthetics.
* Patients with a prior allergic reaction to Morphine and Hydromorphone.
* Patients undergoing any other unrelated surgical procedure to the breast reconstruction.
* Patient refusal to participate.
* Patient required major abdominal surgery within four weeks prior to enrollment.
* Patients being treated for chronic pain or using daily intake of opioid analgesics.
* Patients with a history of abuse of recreational drugs or alcohol.
* Patients with any laboratory values or underlying disease, which in the investigator's opinion would preclude them from participation in the trial, specifically: (A) significant liver dysfunction (eg. bilirubin, AST and/or ALT >1.5 times the upper limit of normal value (B) cardiac conduction defects noted by history or on the pre-op screening EKG.
* Pregnant or breast feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-12; Primary Completion 2006-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Total Postoperative Opioid Use by Patient | Measurements performed and recorded every 6 hours while patient is hospitalized.

CONTACTS AND LOCATIONS:
Overall Officials: Charles E. Butler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org